CLINICAL TRIAL: NCT02240667
Title: Drug Persistence/Adherence in Patients Being Treated With Dabigatran Etexilate or VKA for Stroke Prevention in Non-valvular Atrial Fibrillation (SPAF)
Brief Title: Drug Persistence/Adherence in Patients Treated With Dabigatran or VKA for Stroke Prevention in Non Valvular Atrial Fibrillation (SPAF)
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1160.218
Record Dates: First submitted 2014-09-15; First posted 2014-09-16 (Estimated); Results first posted 2019-04-19 (Actual); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Dabigatran; acarboxyprothrombin; Phenprocoumon

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Subjects with atrial fibrillation
  Interventions: Drug: Dabigatran etexilate; Drug: Vitamin K antagonists

INTERVENTIONS:
Drug: Dabigatran etexilate — 150 mg or 110 mg capsules twice daily
Drug: Vitamin K antagonists — International Normalized Ratio (INR) 2-3
  Other Names: Phenprocoumon

SUMMARY:
1600 AF patients receiving Pradaxa or VKA for stroke prevention will be followed up for 12 months in quarterly visits. Prescriptions, adverse events and (if applicable) reasons for definitive treatment discontinuation will be collected. At 6 months, patient adherence will be assessed, using the Morisky Score.

ELIGIBILITY:
Inclusion criteria:

* Newly prescribed treatment with Pradaxa® (dabigatran etexilate)/VKA in the indication "Stroke prevention in non-valvular atrial fibrillation" (AF) respecting the indication and contraindications as described in the respective Summary of Product Characteristics for Pradaxa® 110 mg or 150 mg hard capsules or the appropriate VKA (patients are eligible for both Pradaxa® and VKA therapy).
* Treatment with dabigatran etexilate or VKA is given in accordance with the respective Summaries of Product Characteristics. The routine diagnostic procedures and treatment that would be undertaken irrespective of the study are unaffected.
* Only patients who are eligible both for therapy with Pradaxa® and for therapy with VKA in accordance with the respective Summaries of Product Characteristics will be documented (patients eligible for VKA and Pradaxa®)
* Patients must have signed the patient consent form prior to inclusion in the Non-Interventional Study (NIS).

Exclusion criteria:

* Patients with the general and special contraindications mentioned in the packaging leaflet or Summary of Product Characteristics must not be included.
* Patients participating at the same time or within the last 30 days in another Non-Interventional Study (NIS) or an interventional clinical trial must not be included.
* Patients treated with anticoagulants for a condition other than non-valvular atrial fibrillation must not be included.
* Pradaxa® and VKA should not be used during pregnancy and lactation. Pregnant or breastfeeding women must therefore not be included in the NIS.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: AF patients
Sampling Method: Probability Sample
Enrollment: 1506 (Actual)
Dates: Start 2014-09-18 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- Multiple Locations, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In this study 1506 patients were entered, 1421 patients had at least one documented prescription of dabigatran etexilate (DE) or vitamin K antagonists (VKA)and were analyzed in the Treated set. 952 patients were matched 1:1 based on Propensity Score (PS).
Pre-assignment Details: The patients were enrolled from 1000 sites from Germany. Approximately 2/3 (about 670) will be community-based primary care internists/general practitioners and approximately 1/3 (about 330) community-based cardiologists across Germany.
Groups:
- Dabigatran (Dabigatran vs VKA): Patients with non-valvular AF treated with Dabigatran as the first Oral Anticoagulants (OACs) for stroke prevention.
- Vitamin K Antagonists (VKA): Patients with non-valvular AF treated with VKA as the first Oral Anticoagulants (OACs) for stroke prevention.
Period: Overall Study
Arm/Group | Dabigatran (Dabigatran vs VKA) | Vitamin K Antagonists (VKA)
Started | 771 | 650
Completed | 771 | 650
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Treated set (TS) includes all patients with main diagnosis of nonvalvular AF (=IC 2) with at least one evaluable efficacy endpoint (being on treatment is an efficacy endpoint).
Groups:
- Total: Total of all reporting groups
Arm/Group | Dabigatran (Dabigatran vs VKA) | Vitamin K Antagonists (VKA) | Total
Number analyzed (Participants) | 771 | 650 | 1421
Age, Continuous [Median (Full Range); unit: Years] — Population: TS
  Years
    Overall | 75 [23 to 96] | 75 [38 to 96] | 75 [23 to 96]
    Dabigatran vs VKA(matched pop): number analyzed (Participants) | 476 | 476 | 952
    Dabigatran vs VKA(matched pop) | 75 [40 to 96] | 75 [38 to 96] | 75 [38 to 96]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: TS
  Participants
    Overall: Female | 339 | 284 | 623
    Overall: Male | 432 | 366 | 798
    Dabigatran vs VKA(matched pop): number analyzed (Participants) | 476 | 476 | 952
    Dabigatran vs VKA(matched pop): Female | 214 | 205 | 419
    Dabigatran vs VKA(matched pop): Male | 262 | 271 | 533
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Race and Ethnicity was not reported in this trial Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Treated With Anticoagulation Initially Started at the 12 Month
Description: Percentage of patients treated with the initially allocated anticoagulant at the 12-month visit, defined as Kaplan Meier estimate at 12 months for persistence, stratified for dabigatran etexilate and VKA.Persistence is defined as the time between initiation and permanent discontinuation of therapy. The initiation date is the documented start of treatment (at visit 1), and the date of permanent discontinuation is the documented permanent discontinuation of dabigatran etexilate or VKA therapy.
Time Frame: 12 month (Visit 5)
Population: Patients in the TS who were matched 1:1 based on propensity score matching in order to ensure comparability of outcome variables between both treatment groups (dabigatran etexilate and VKA).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Dabigatran (Dabigatran vs VKA): Patients with non-valvular AF treated with dabigatran as the first Oral Anticoagulants (OACs) were matched 1:1 based on Propensity Score (PS).
- VKA (Dabigatran vs VKA): Patients with non-valvular AF treated with VKA as the first Oral Anticoagulants (OACs) were matched 1:1 based on Propensity Score (PS).
Arm/Group | Dabigatran (Dabigatran vs VKA) | VKA (Dabigatran vs VKA)
Number analyzed (Participants) | 476 | 476
percentage of participants | 89.5 [86.3 to 91.9] | 89.5 [86.3 to 92.0]
Statistical Analysis 1: Comparison: Dabigatran (Dabigatran vs VKA) vs VKA (Dabigatran vs VKA); Persistence in both treatment groups was compared by means of the stratified Log-rank test; Test type: Other; p = 0.8496, stratified log-rank test

2. Secondary Outcome: Percentage of Patients With Low, Medium or High Adherence at the Timepoint of 6 Months-visit.
Description: Percentage of patients with low, medium or high adherence at the 6-month visit, stratified for dabigatran etexilate and VKA; categorisation is done on the basis of the Morisky questionnaire (high, medium and low adherence with a Morisky score of 0, 1 to 2, and > 2, respectively).
Time Frame: 6 month (visit 3)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Dabigatran (Dabigatran vs VKA) | VKA (Dabigatran vs VKA)
Number analyzed (Participants) | 476 | 476
Percentage of participants
  Low | 19.12 | 23.74
  Medium | 45.8 | 46.85
  High | 5.88 | 3.99
  Missing | 29.2 | 25.42

3. Secondary Outcome: Number of Patients With the Reason for Definitive Treatment Discontinuation
Description: Number of patients with the reason for definitive treatment discontinuation
Time Frame: Visit 2, 3, 4 and 5 (after approx. 3, 6, 9 and 12 months of treatment)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Dabigatran (Dabigatran vs VKA) | VKA (Dabigatran vs VKA)
Number analyzed (Participants) | 476 | 476
Participants
  Visit 2 (Month 3): number analyzed (Participants) | 2 | 2
  Visit 2 (Month 3): Serious adverse event | 0 | 0
  Visit 2 (Month 3): Patient's wish | 1 | 1
  Visit 2 (Month 3): Decision of physician | 1 | 0
  Visit 2 (Month 3): Other | 0 | 1
  Visit 3 (Month 6): number analyzed (Participants) | 3 | 4
  Visit 3 (Month 6): Serious adverse event | 1 | 1
  Visit 3 (Month 6): Patient's wish | 0 | 1
  Visit 3 (Month 6): Decision of physician | 1 | 1
  Visit 3 (Month 6): Other | 1 | 1
  Visit 4 (Month 9): number analyzed (Participants) | 0 | 3
  Visit 4 (Month 9): Serious adverse event | 0 | 0
  Visit 4 (Month 9): Patient's wish | 0 | 0
  Visit 4 (Month 9): Decision of physician | 0 | 2
  Visit 4 (Month 9): Other | 0 | 1
  Visit 5 (Month 12): number analyzed (Participants) | 3 | 2
  Visit 5 (Month 12): Serious adverse event | 0 | 0
  Visit 5 (Month 12): Patient's wish | 1 | 0
  Visit 5 (Month 12): Decision of physician | 0 | 2
  Visit 5 (Month 12): Other | 2 | 0

ADVERSE EVENTS:
Time Frame: From start of treatment until six days after permanent treatment discontinuation or end of study, up to 12 months.
Description: The Treated set (TS) includes all patients with main diagnosis of nonvalvular AF with at least one evaluable efficacy endpoint (being on treatment is an efficacy endpoint). Treatment emergent Adverse events were reported.
Arm/Group | Dabigatran (Dabigatran vs VKA) | Vitamin K Antagonists (VKA)
All-Cause Mortality (participants affected / at risk) | 10/771 | 5/650
Serious Adverse Events (participants affected / at risk) | 45/771 | 39/650
Other Adverse Events (participants affected / at risk) | 0/771 | 0/650
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dabigatran (Dabigatran vs VKA) (N=771) | Vitamin K Antagonists (VKA) (N=650)
Cardiac failure (Cardiac disorders) | 4 | 5
Atrial fibrillation (Cardiac disorders) | 2 | 3
Acute coronary syndrome (Cardiac disorders) | 1 | 4
Cardiac arrest (Cardiac disorders) | 1 | 3
Angina pectoris (Cardiac disorders) | 1 | 2
Myocardial infarction (Cardiac disorders) | 2 | 1
Ventricular fibrillation (Cardiac disorders) | 2 | 0
Atrial tachycardia (Cardiac disorders) | 1 | 0
Mitral valve disease (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 2 | 0
Optic ischaemic neuropathy (Eye disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 1
Ileus (Gastrointestinal disorders) | 1 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 1
Oesophageal ulcer (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Large intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 1 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Duodenal perforation (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Anal haemorrhage (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Papilla of Vater stenosis (Gastrointestinal disorders) | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 1 | 0
Generalised oedema (General disorders) | 1 | 0
Cholestasis (Hepatobiliary disorders) | 0 | 1
Jaundice (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 1
Sepsis (Infections and infestations) | 3 | 0
Lung infection (Infections and infestations) | 2 | 1
Wound infection (Infections and infestations) | 1 | 1
Bronchitis (Infections and infestations) | 1 | 1
Paronychia (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Biliary tract infection (Infections and infestations) | 0 | 1
Peritonitis (Infections and infestations) | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Wound complication (Injury, poisoning and procedural complications) | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 1
Electrocardiogram change (Investigations) | 0 | 1
Troponin I increased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 1 | 1
Cerebrovascular accident (Nervous system disorders) | 2 | 0
Syncope (Nervous system disorders) | 2 | 0
Cerebral microangiopathy (Nervous system disorders) | 1 | 0
Chorea (Nervous system disorders) | 1 | 0
Dysarthria (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Restlessness (Psychiatric disorders) | 1 | 0
Chronic kidney disease (Renal and urinary disorders) | 2 | 1
Haematuria (Renal and urinary disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Mediastinal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haematoma (Vascular disorders) | 1 | 0
Embolism (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
Hypertensive crisis (Vascular disorders) | 0 | 1
Aortic dissection (Vascular disorders) | 0 | 1
Peripheral ischaemia (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2016-01-04): https://cdn.clinicaltrials.gov/large-docs/67/NCT02240667/Prot_000.pdf
  • Statistical Analysis Plan (2015-08-13): https://cdn.clinicaltrials.gov/large-docs/67/NCT02240667/SAP_001.pdf